CLINICAL TRIAL: NCT00290238
Title: Percutaneous Neuromodulation Therapy With Chronic Low Back Pain Patients With or Without Lower Extremity Pain - A Randomized, Controlled, Parallel Groups Study
Brief Title: Percutaneous Neuromodulation Therapy (PNT) With Chronic Low Back Pain Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow recruitment and high dropout rates
Sponsor: RS Medical (Industry)
Responsible Party: Vice President of Research and Development, RS Medical
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RSMED-K011702-PNT02
Record Dates: First submitted 2006-02-08; First posted 2006-02-10 (Estimated); Results first posted 2009-03-09 (Estimated); Last update posted 2009-06-01 (Estimated); Status verified 2009-05

CONDITIONS: Low Back Pain
Keywords: Chronic Low Back Pain; Lower Extremity Pain; Central Sensitization; Percutaneous Neuromodulation Therapy
MeSH Terms: conditions — Low Back Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PNT (Experimental)
  Interventions: Device: Vertis Percutaneous Neuromodulation Therapy (PNT)
- TENS (Sham Comparator)
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)

INTERVENTIONS:
Device: Vertis Percutaneous Neuromodulation Therapy (PNT) — * Ten PNT sessions in eleven weeks
  * On average, one PNT session per week
  * Ten lumbar Safeguide electrodes (three centimeters in length) deployed per lumbar montage
  * Forty-five minutes of electrical stimulation for each session
  * Electrical stimulation parameters:
    * Continuous 50 Hz current
    * Charge-balanced, biphasic (each phase is 200 microsec), rectangular waveform
    * Intensity to subject's tolerance for ten minutes then increased to a mildly uncomfortable level
  Other Names: PNT; Vertis
  Arms: PNT
Device: Transcutaneous Electrical Nerve Stimulation (TENS) — * Ten TENS sessions in eleven weeks
  * On average, one TENS session per week
  * Four 2-inch (5.1 centimeters) diameter pads applied per TENS lumbar montage
  * Forty-five minutes of electrical stimulation for each session
  * Electrical stimulation parameters:
    * Current at 2 Hz-low frequency
    * Pulse trains delivered as asymmetric, biphasic, square waveform current, with pulse width lasting 20 microsec
    * Intensity titrated according to subject's sensory threshold
    * To maintain blinding, the treating physician or clinician will check on the subject after 10 minutes and dial the channels down just prior to the point of turning off the device.
  Other Names: TENS; Transcutaneous electrical nerve stimulation; surface stimulation
  Arms: TENS

SUMMARY:
The purpose of this study is to assess the benefits of Percutaneous Neuromodulation Therapy when compared to a reference sham treatment in the treatment of patients who have undergone surgical intervention for chronic low back pain with or without a radiating lower extremity pain component.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain for at least 6 months
* If lower extremity pain present, must be present for at least 3 months
* Visual analog scale (VAS) score for low back pain at least 50 out of 100
* Lumbar or lumbosacral surgical intervention without pain relief
* Central sensitization symptoms
* Agrees to follow randomized treatment plan
* 18 years of age or older
* Signed informed consent form

Exclusion Criteria:

* Significant change to low back or lower extremity pain within 4 weeks prior to enrollment
* Nociceptive and/or neuropathic pain symptoms in the spine due to structural and/or mechanical instabilities
* Three or more lumbar or lumbosacral surgical interventions; one or more surgical interventions in areas other than lumbar or lumbosacral spine
* Three or more lumbar vertebral segments fused
* Lumbar or lumbosacral surgical intervention in last 9 months; areas other than lumbar or lumbosacral in last 12 months
* Any additional surgical intervention required 3 months post-enrollment
* Symptoms consistent with sympathetically-maintained pain
* Evidence of serious neurological deficits or impairments
* Significant changes in pain medications within 4 weeks prior to enrollment
* Psychosocial issues that conflict with valid reporting by patient
* Prior treatment with percutaneous electrical stimulation or sensitivity to electrical stimulation
* Current use of another electrical stimulation device for low back or lower extremity pain
* Current enrollment in another clinical trial within the last 30 days
* Current or prior malignancy or cancer
* Serious or uncontrolled systemic illness
* Body mass index (BMI) greater than 40
* Pregnant or intends to become pregnant during the study
* Implanted medical device
* Relationship with study staff
* Unable to attend study office visits or complete study measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2005-12; Primary Completion 2007-11 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Carroll, Study Director — RS Medical
Locations (8):
- United States (8):
  - UCSD Pain Research Center, La Jolla, California
  - Center for Prospective Outcome Studies, Atlanta, Georgia
  - Mossberg Research Group, Eugene, Oregon
  - Pain Specialists of Southern Oregon, Medford, Oregon
  - Neuropsychiatric Pain Medicine Association of Tennessee, Knoxville, Tennessee
  - Physical Medicine & Rehabilitation Center, Seymour, Tennessee
  - Texas Back Institute - Denton, Denton, Texas
  - Texas Back Institute CRO, Plano, Texas

REFERENCES:
- [Background] White PF, Ghoname EA, Ahmed HE, Hamza MA, Craig WF, Vakharia AS. The effect of montage on the analgesic response to percutaneous neuromodulation therapy. Anesth Analg. 2001 Feb;92(2):483-7. doi: 10.1097/00000539-200102000-00038. PMID 11159255
- [Background] Ghoname ES, Craig WF, White PF, Ahmed HE, Hamza MA, Gajraj NM, Vakharia AS, Noe CE. The effect of stimulus frequency on the analgesic response to percutaneous electrical nerve stimulation in patients with chronic low back pain. Anesth Analg. 1999 Apr;88(4):841-6. doi: 10.1097/00000539-199904000-00030. PMID 10195535
- [Background] White PF, Craig WF, Vakharia AS, Ghoname E, Ahmed HE, Hamza MA. Percutaneous neuromodulation therapy: does the location of electrical stimulation effect the acute analgesic response? Anesth Analg. 2000 Oct;91(4):949-54. doi: 10.1097/00000539-200010000-00034. PMID 11004055
- [Background] Borg-Stein J, Seroussi RE, Gomba L, Meleger A, Schmitt S, Leep E, Glassman JH, Revord J, Condon J, Bensen E, Fitzthum JE, Fowler BC, Gliner BE, Firlik AD. Safety and efficacy of percutaneous neuromodulation therapy in the management of subacute radiating low back pain. Pain Pract. 2003 Jun;3(2):125-34. doi: 10.1046/j.1533-2500.2003.03019.x. PMID 17163911

RESULTS

PARTICIPANT FLOW:
Groups:
- Percutaneous Neuromodulation Therapy (PNT): Active/test group receiving 10 Percutaneous Neuromodulation Therapy (PNT) sessions of 45 minutes each over 11 weeks. PNT delivers 50 Hz current in a charge-balanced, biphasic, rectangular waveform.
- Transcutaneous Electrical Nerve Stimulation (TENS): Sham comparator group receiving 10 TENS sessions of 45 minutes each over 11 weeks. Delivered 2 Hz pulse trains as asymmetric, biphasic, square waves with pulse width of 20 microseconds.
Period: Overall Study
Arm/Group | Percutaneous Neuromodulation Therapy (PNT) | Transcutaneous Electrical Nerve Stimulation (TENS)
Started | 57 | 65 (One subject had an invalid birth date and was excluded from the Age Categorical counts.)
Completed | 15 | 24
Not Completed | 42 | 41
Not completed — Study terminated | 27 | 27
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 15 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Percutaneous Neuromodulation Therapy (PNT) | Transcutaneous Electrical Nerve Stimulation (TENS) | Total
Number analyzed (Participants) | 57 | 65 | 122
Age Categorical [Number; unit: participants] — One subject had an invalid birth date and was excluded from the Age Categorical counts.
  participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 43 | 54 | 97
    >=65 years | 14 | 10 | 24
Age Continuous [Mean (Standard Deviation); unit: years] | 53.7 (15.1) | 55.9 (11.0) | 54.8 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 37 | 70
  Male | 24 | 28 | 52
Region of Enrollment [Number; unit: participants]
  United States | 57 | 65 | 122

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Time-averaged Pain Intensity Visual Analog Scale (VAS) Score
Description: Visual analog scale (VAS) for pain (100mm line with "0/No pain" on the left and "100/Worst pain imaginable" on the right). Subjects drew vertical line to indicate pain. Time-averaged method accounts for time between visits by dividing area beneath the score curve by time between first and last available visits.
Time Frame: Time-averaged from the first available observation to the last available observation (12 months for completed subjects)
Population: Analysis population was intention to treat (ITT), excluding subjects who had no follow-up (after the initial 10-week treatment phase) data available.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Percutaneous Neuromodulation Therapy (PNT) | Transcutaneous Electrical Nerve Stimulation (TENS)
Number analyzed (Participants) | 51 | 64
mm
  Back pain | -10.9 (3.1) [29.5 to 89.5] | -11.7 (2.7) [35.5 to 88.5]
  Radiating leg/buttock pain | -12.8 (3.2) | -9.8 (2.9)

2. Secondary Outcome: Total Expenditure Per Day on All Lower Back Pain Related Interventions
Description: Expenditures were assessed by patient report at each visit. Interventions were coded to Current Procedural Terminology (CPT) 2008; costs were derived from Medicare, Managed Care, and Workers' Comp fees. Costs for providers assume 30 minutes at returning patient rate. Drug costs were coded to a dictionary extrapolated from 2008 market prices.
Time Frame: Baseline, Month 01, Month 02, Month 04, Month 06, Month 08, Month 10, Month 12
Population: Analysis population was intention to treat (ITT).
Measure: Median (Full Range); unit: Dollars
Arm/Group | Percutaneous Neuromodulation Therapy (PNT) | Transcutaneous Electrical Nerve Stimulation (TENS)
Number analyzed (Participants) | 57 | 65
Dollars | 2.97 [0 to 77.20] | 5.30 [0 to 118.08]

ADVERSE EVENTS:
Arm/Group | Percutaneous Neuromodulation Therapy (PNT) | Transcutaneous Electrical Nerve Stimulation (TENS)
Serious Adverse Events (participants affected / at risk) | 3 | 3
Other Adverse Events (participants affected / at risk) | 29 | 38
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Percutaneous Neuromodulation Therapy (PNT) | Transcutaneous Electrical Nerve Stimulation (TENS)
Bruise/abrasion/fracture/other injury (Injury, poisoning and procedural complications) | 1/57 (1) | 0/65 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1/57 (1) | 0/65 (0)
Surgery (Musculoskeletal and connective tissue disorders) | 1/57 (1) | 0/65 (0)
Myocardial infarction (Cardiac disorders) | 0/57 (0) | 1/65 (1)
Low back pain (serious events) (Musculoskeletal and connective tissue disorders) | 0/57 (0) | 2/65 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Percutaneous Neuromodulation Therapy (PNT) | Transcutaneous Electrical Nerve Stimulation (TENS)
Low back pain (non-serious events) (Musculoskeletal and connective tissue disorders) | 17/57 (44) | 22/65 (57)
Leg/buttock/hip or radiating pain (Musculoskeletal and connective tissue disorders) | 7/57 (9) | 9/65 (12)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2/57 (2) | 7/65 (8)
Arm/shoulder pain (Musculoskeletal and connective tissue disorders) | 2/57 (2) | 5/65 (6)
Bruise/abrasion/fracture/other injury (Injury, poisoning and procedural complications) | 3/57 (3) | 7/65 (8)
Headache (General disorders) | 2/57 (3) | 4/65 (6)
Drug reaction (Injury, poisoning and procedural complications) | 1/57 (3) | 4/65 (4)
Virus (Infections and infestations) | 2/57 (3) | 3/65 (5)
Urinary/bladder infection (Infections and infestations) | 4/57 (4) | 0/65 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If the PI expects to participate in the publication or presentation of data generated in the performance of the study, any reports, abstracts, manuscripts, or other presentation materials shall be submitted to the sponsor for review prior to submission for publication or presentation. The sponsor shall have 30 calendar days to respond with any requested revisions in order to protect the sponsor's confidential information.